CLINICAL TRIAL: NCT01280123
Title: A Multi-Center, Double-Blind, Placebo-Controlled Phase II Study of Pioglitazone in Early Parkinson's Disease
Brief Title: Pioglitazone in Early Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FS-ZONE; 5U01NS043128-12 (NIH)
Record Dates: First submitted 2010-12-03; First posted 2011-01-20 (Estimated); Results first posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2013-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Biomarkers
MeSH Terms: conditions — Parkinson Disease | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 15 mg pioglitazone (Experimental): 15 mg pioglitazone
  Interventions: Drug: Pioglitazone
- 45 mg pioglitazone (Experimental): 45 mg pioglitazone
  Interventions: Drug: Pioglitazone
- Matching Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pioglitazone — Oral capsules of Pioglitazone (15 mg capsules) either 15 mg/qd or 45 mg/qd
  Subjects will titrate in a blinded fashion to 30 mg/day after 2 weeks and to 45 mg per day) 2 weeks later as tolerated.
  Other Names: Pioglitazone Hydrochloride; ACTOS (R)
  Arms: 15 mg pioglitazone; 45 mg pioglitazone
Drug: placebo — Placebo will contain microcrystalline cellulose. An over-encapsulation process will be conducted in accordance with Clinical Good Manufacturing Procedures (cGMP) regulations to create a dosage form for the active study drug that will be indistinguishable from the comparator (Placebo) capsule.
  Arms: Matching Placebo

SUMMARY:
This is a multi-center, double-blind, placebo controlled clinical trial of two dosages of oral pioglitazone (15 milligram(mg) and 45 milligram (mg)) for safety, tolerability, and futility.

Subjects who are on stable dose of rasagiline 1 mg/day or selegiline 10 mg/day for at least 8 weeks but no more than 8 months, will be randomized to one of two dosages of oral pioglitazone (15 mg and 45 mg) or matching placebo.

The study will measure disease progression by the change in total Unified Parkinson's Disease Rating Scale (UPDRS) score between the baseline visit and 44 weeks.

DETAILED DESCRIPTION:
A Multi-Center, Double-Blind, Placebo-Controlled Phase II Study of Pioglitazone in Early Parkinson's Disease (PD). The patient population has early stage PD (< 5 years from diagnosis), must be treated with 1 mg/day of rasagiline or 10 mg/day of selegiline for at least 8 weeks but not more than 8 months prior to enrollment.

The primary objective of this clinical trial is to assess the futility of pioglitazone on PD disease progression as measured by the change in total UPDRS score between the baseline visit and 44 weeks. The secondary objectives of the study are to collect additional efficacy and safety/tolerability data to be used in planning a subsequent Phase III trial of pioglitazone in early, treated PD. Measures of cognition, mood and blood- and urine-based biomarkers will also be explored. Subjects in this trial are randomly assigned in a 1:1:1 ratio to one of three study arms: 15 mg, 45 mg or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent.
2. Men and women with idiopathic PD of less than 5 years duration from diagnosis with a Hoehn and Yahr Stage < 2.
3. On stable dosage of rasagiline 1 mg/day or selegiline 10 mg/day for at least 8 weeks but not more than 8 months prior to baseline. Expected to remain on stable dose of rasagiline or selegiline as the only treatment for their PD for the duration of the study (44 weeks).
4. Diagnosis must be confirmed by bradykinesia plus one of the other cardinal signs (resting tremor, rigidity) being present, without any other known or suspected cause of parkinsonism. The clinical signs must be asymmetric.
5. Subjects may be taking stable doses (30 days) of anticholinergics or creatine (< 5gm/day) but must be expected to remain on the same dose.
6. Age > 30 years.
7. Women who are not postmenopausal or surgically sterile must use a medically accepted contraceptive regimen for at least 60 days before the baseline visit, and agree to continue such use throughout the duration of the study and for 30 days after the final dose of study drug.

Exclusion Criteria:

1. Exposure to dopaminergic PD therapy or amantadine within 60 days prior to baseline visit or for 90 days or more at any point in the past
2. Use of any of the following drugs within 180 days prior to baseline: neuroleptics, metoclopramide, alpha-methyldopa, clozapine, olanzapine and flunarizine.
3. Use of any of the following drugs within 90 days prior to baseline: methylphenidate, cinnarizine, reserpine, tetrabenazine, amphetamine or monoamine oxidase (MAO)-A inhibitors (pargyline, phenelzine, and tranylcypromine).
4. Presence of drug-induced parkinsonism (e.g., metoclopramide, flunarizine), metabolic identified neurogenetic disorders (e.g., Wilson's disease), encephalitis, or other atypical Parkinsonian syndromes (e.g., progressive supranuclear palsy, multiple system atrophy).
5. Participation in other drug studies or receipt of other investigational drugs within 30 days prior to baseline or during the study.
6. Presence of freezing.
7. Any clinically significant psychiatric or medical condition or laboratory abnormality, which would in the judgment of the Investigator interfere with the subject's ability to participate.
8. History of stereotaxic brain surgery for PD
9. Clinically significant structural brain disease that the investigator believes would interfere with study evaluations.
10. History of congestive heart failure.
11. Use of pioglitazone or rosiglitazone within 90 days before randomization.
12. Known intolerance to pioglitazone or rosiglitazone.
13. Allergy to rasagiline or selegiline, or contraindication to rasagiline or selegiline use.
14. Type I or Type II diabetes mellitus.
15. HgbA1C greater than or equal to 6% at Screening.
16. Known liver disease or elevation of AST or ALT greater than 2.5 times the upper limit of normal.
17. Known history of osteoporosis. All women ≥ 65 years of age or men and woman at high risk of osteoporosis should have documented evidence of screening for osteoporosis. Factors associated with high risk of osteoporosis include: previous non traumatic fracture, chronic glucocorticoid use, body weight under 58 kg, family history of hip fracture, current cigarette smoking, and excessive alcohol intake.
18. Drug or alcohol use or dependence that, in the opinion of the Investigator, would interfere with the safe conduct of the study.
19. Significant peripheral edema (2+ or more) of the extremities of any etiology.
20. Current or planned use of gemfibrozil or rifampin during the trial.
21. History of bladder cancer.
22. Evidence of hematuria which has not been evaluated for evidence of bladder cancer. (Documentation of work up or a repeat urine test that was negative for hematuria and the primary care physician or urologist does not feel that further work up is required.)
23. History of macular edema.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Simuni, MD, Study Director — Northwestern University; Karl Kieburtz, MD MPH, Study Director — University of Rochester
Locations (38):
- United States (38):
  - Univeristy of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - The Parkinson's & Movement Disorder Institute, Fountain Valley, California
  - University of Southern California, Los Angeles, California
  - University of California San Fransisco, San Francisco, California
  - Univeristy of Colorado Denver, Aurora, Colorado
  - University of Florida, Gainsville, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Pacific Health Research & Education Institute, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - LSU Health Science Center Shreveport, Shreveport, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - Washington University, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - SUNY Downstate Medical Center, Brooklyn, New York
  - North Shore - LIJ Health System, Manhasset, New York
  - Duke University, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Result] NINDS Exploratory Trials in Parkinson Disease (NET-PD) FS-ZONE Investigators. Pioglitazone in early Parkinson's disease: a phase 2, multicentre, double-blind, randomised trial. Lancet Neurol. 2015 Aug;14(8):795-803. doi: 10.1016/S1474-4422(15)00144-1. Epub 2015 Jun 23. PMID 26116315
- [Derived] Carta AR, Simuni T. Thiazolidinediones under preclinical and early clinical development for the treatment of Parkinson's disease. Expert Opin Investig Drugs. 2015 Feb;24(2):219-27. doi: 10.1517/13543784.2015.963195. Epub 2014 Sep 17. PMID 25227476

RESULTS

PARTICIPANT FLOW:
Groups:
- 15 mg Pioglitazone: 15 mg pioglitazone
  Pioglitazone: Oral capsules of Pioglitazone (15 mg capsules) either 15 mg/qd or 45 mg/qd or matching placebo
  44 weeks: Subjects who are on stable dose of rasagiline 1 mg/day or selegiline 10 mg/day, for at least 8 weeks but no more than 8 months, will begin randomized dose of study drug. Subjects will titrate in a blinded fashion to 30 mg/day after 2 weeks and to 45 mg per day) 2 weeks later as tolerated. Subjects will be followed on study drug for 44 weeks.
- 45 mg Pioglitazone: 45 mg pioglitazone
  Pioglitazone: Oral capsules of Pioglitazone (15 mg capsules) either 15 mg/qd or 45 mg/qd or matching placebo
  44 weeks: Subjects who are on stable dose of rasagiline 1 mg/day or selegiline 10 mg/day, for at least 8 weeks but no more than 8 months, will begin randomized dose of study drug. Subjects will titrate in a blinded fashion to 30 mg/day after 2 weeks and to 45 mg per day) 2 weeks later as tolerated. Subjects will be followed on study drug for 44 weeks.
Period: Overall Study
Arm/Group | 15 mg Pioglitazone | 45 mg Pioglitazone | Matching Placebo
Started | 72 | 67 | 71
Completed | 71 | 63 | 70
Not Completed | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 mg Pioglitazone | 45 mg Pioglitazone | Matching Placebo | Total
Number analyzed (Participants) | 72 | 67 | 71 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.6) | 58.8 (9.2) | 59.0 (9.9) | 59.7 (9.9)
Sex/Gender, Customized [Number; unit: participants]
  Males | 53 | 47 | 48 | 148
  Females | 19 | 20 | 23 | 62
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Latino whites | 58 | 63 | 63 | 184
  Racial/Ethnic Minority | 14 | 4 | 8 | 26
Years of education [Mean (Standard Deviation); unit: years] | 17.1 (3.1) | 16.2 (3.3) | 16.8 (3.0) | 16.7 (3.1)
Right-handed [Number; unit: participants]
  Yes | 62 | 62 | 62 | 186
  No | 10 | 5 | 9 | 24
Duration of PD symptoms (years) [Mean (Standard Deviation); unit: years] | 2.3 (1.9) | 2.0 (1.2) | 2.3 (2.3) | 2.2 (1.9)
Time since PD diagnosis (years) [Mean (Standard Deviation); unit: years] | 0.8 (0.7) | 0.7 (0.7) | 0.8 (0.7) | 0.7 (0.7)
Total Unified Parkinson's Disease Rating Scale (UPDRS) [Mean (Standard Deviation); unit: units on a scale] — The Total UPDRS is the sum of parts I, II, and III. The possible range of the total UPDRS is from 0-176. Higher values indicate worse outcomes.
  units on a scale | 23.8 (9.9) | 21.2 (8.8) | 21.7 (8.7) | 22.2 (9.2)
UPDRS mental [Mean (Standard Deviation); unit: units on a scale] — The UPDRS mental score is the sum of the questions in part I. The possible range of the UPDRS mental is from 0-16. Higher values indicate worse outcomes.
  units on a scale | 0.8 (0.9) | 0.8 (0.9) | 0.9 (1.1) | 0.8 (1.0)
UPDRS motor [Mean (Standard Deviation); unit: units on a scale] — The UPDRS motor score is the sum of the questions in part III. The possible range of the UPDRS motor is from 0-108. Higher values indicate worse outcomes.
  units on a scale | 17.7 (7.7) | 15.0 (7.1) | 15.3 (6.5) | 15.8 (7.1)
UPDRS ADL [Mean (Standard Deviation); unit: units on a scale] — The UPDRS ADL score is the sum of the questions in part II (activities of daily living). The possible range of the UPDRS ADL is from 0-52. Higher values indicate worse outcomes.
  units on a scale | 5.9 (3.2) | 5.5 (2.9) | 5.5 (3.0) | 5.6 (3.0)
Ambulatory capacity [Mean (Standard Deviation); unit: units on a scale] — Ambulatory Capacity is calculated as the sum of items 13-15, 29, 30 of the Unified Parkinson's Disease Rating Scale (UPDRS). It ranges from 0-20. Higher scores are worse.
  units on a scale | 1.1 (0.9) | 0.8 (0.8) | 1.1 (0.9) | 1.0 (0.9)
Schwab and England Activities of Daily Living scale (SEADL) [Mean (Standard Deviation); unit: units on a scale] — The modified Schwab and England Activities of Daily Living is a single question ranging from 0-100% with anchors for each 10% interval. Higher scores are better (100% completely independent- 0% vegetative).
  units on a scale | 93.8 (4.9) | 94.1 (5.0) | 93.9 (5.0) | 93.9 (4.9)
Parkinson's Disease Questionnaire 39 (PDQ-39) Summary Index [Mean (Standard Deviation); unit: units on a scale] — The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality. The total score ranges from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better quality of life.
  units on a scale | 8.5 (8.1) | 8.1 (5.9) | 10.6 (7.9) | 9.1 (7.4)
Geriatric Depression Scale (GDS) [Mean (Standard Deviation); unit: units on a scale] — Short version. 15 questions. A score of 0 to 5 is normal. A score greater than 5 suggests depression.
  units on a scale | 1.4 (1.4) | 1.1 (1.3) | 1.8 (1.9) | 1.4 (1.6)
Mattis-Dementia Rating scale [Mean (Standard Deviation); unit: units on a scale] — Mattis Dementia Rating scale (DRS-2) raw score is the sum of 5 raw sub-scores (attention has possible 37 points, initiation/perseveration has possible 37 points, construction has possible 6 points, conceptualization has possible 39 points, memory has possible 25 points). Total range is 0-144. Higher scores are better.
  units on a scale | 138.6 (8.2) | 138.8 (10.2) | 138 (11.4) | 138.4 (9.9)
rasagiline/selegiline use [Number; unit: participants] — Proportion of patients on stable regimen of either 1 mg/day rasagiline or 10 mg/day selegiline at baseline.
  participants
    rasagiline use | 60 | 57 | 60 | 177
    selegiline use | 12 | 10 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Unified Parkinson's Disease Rating Scale (UPDRS) Score From Baseline to 44 Weeks
Description: Change in total UPDRS score from baseline to 44 weeks (in subjects treated with rasagiline 1 mg/day or selegiline 10 mg/day).
  The Total UPDRS is the sum of parts I, II, and III. The possible range of the total UPDRS is from 0-176. Higher values indicate worse outcomes.
  The change is 44 weeks - baseline.
Time Frame: 44 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 15 mg Pioglitazone | 45 mg Pioglitazone | Matching Placebo
Number analyzed (Participants) | 72 | 67 | 71
units on a scale | 4.42 (0.95) | 5.13 (0.99) | 6.25 (0.96)

2. Secondary Outcome: Change in Ambulatory Capacity From Baseline to 44 Weeks
Description: This is the sum of the 5 UPDRS questions regarding ambulatory capacity: falling, freezing, walking, gait, postural stability.
  Ambulatory Capacity is calculated as the sum of items 13-15, 29, 30 of the Unified Parkinson's Disease Rating Scale (UPDRS). It ranges from 0-20. Higher scores are worse. Change is 44 weeks - baseline.
Time Frame: 44 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 15 mg Pioglitazone | 45 mg Pioglitazone | Matching Placebo
Number analyzed (Participants) | 72 | 67 | 71
units on a scale | 0.39 [0.16 to 0.61] | 0.38 [0.07 to 0.70] | 0.4 [0.17 to 0.64]

3. Secondary Outcome: Change in Schwab and England Scale From Baseline to 44 Weeks
Description: The modified Schwab and England Activities of Daily Living is a single question ranging from 0-100% with anchors for each 10% interval. Higher scores are better (100% completely independent- 0% vegetative).
Time Frame: 44 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 15 mg Pioglitazone | 45 mg Pioglitazone | Matching Placebo
Number analyzed (Participants) | 72 | 67 | 71
units on a scale | -2.12 [-3.47 to -0.78] | -2.52 [-3.95 to -1.09] | -1.84 [-3.49 to -0.18]

4. Secondary Outcome: Change in Parkinson's Disease Questionnaire (PDQ-39) From Baseline to 44 Weeks
Description: The Parkinson's Disease Questionnaire (PDQ-39) is a short, 39 item measure of quality of life in subjects with Parkinson's disease. The questionnaire covers 8 aspects of quality of life: mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication and bodily discomfort.
  The total score ranges from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better quality of life.
Time Frame: 44 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 15 mg Pioglitazone | 45 mg Pioglitazone | Matching Placebo
Number analyzed (Participants) | 72 | 67 | 71
units on a scale | 2.03 [0.47 to 3.59] | 2.08 [0.32 to 3.84] | 0.08 [-1.59 to 1.76]

5. Secondary Outcome: Change in the Mattis Dementia Rating Scale (DRS-2)From Baseline to 44 Weeks
Description: The Mattis dementia rating scale is a psychometric instrument designed to assess the extent and nature of dementia. Mattis Dementia Rating scale (DRS-2) raw score is the sum of 5 raw sub-scores (attention has possible 37 points, initiation/perseveration has possible 37 points, construction has possible 6 points, conceptualization has possible 39 points, memory has possible 25 points). Total range is 0-144. Higher scores are better.
Time Frame: 44 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 15 mg Pioglitazone | 45 mg Pioglitazone | Matching Placebo
Number analyzed (Participants) | 72 | 67 | 71
units on a scale | 1.16 [-1.26 to 3.58] | 2.11 [-0.41 to 4.63] | 3.16 [0.66 to 5.65]

6. Secondary Outcome: Change in the 15-item Geriatric Depression Scale (GDS-15)From Baseline to 44 Weeks
Description: The Geriatric Depression Scale - 15 is a short 15 yes or no question instrument for assessing depression in the elderly. It has been found to be particularly useful in assessing depression in Parkinson's Disease. A score of 0 to 5 is normal. A score greater than 5 suggests depression.
Time Frame: 44 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 15 mg Pioglitazone | 45 mg Pioglitazone | Matching Placebo
Number analyzed (Participants) | 72 | 67 | 71
units on a scale | 0.13 [-0.33 to 0.58] | 0.38 [-0.10 to 0.85] | 0.18 [-0.37 to 0.72]

ADVERSE EVENTS:
Time Frame: All events during study period (defined as from signing consent to conclusion of study participation 44 weeks).
Description: Adverse event data was elicited by asking an open ended question "What unusual symptoms or medical problems have you experienced since the last visit?"
Arm/Group | 15 mg Pioglitazone | 45 mg Pioglitazone | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 6/72 | 9/67 | 3/71
Other Adverse Events (participants affected / at risk) | 63/72 | 51/67 | 59/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg Pioglitazone (N=72) | 45 mg Pioglitazone (N=67) | Matching Placebo (N=71)
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Transient ischemic attack (Nervous system disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 15 mg Pioglitazone (N=72) | 45 mg Pioglitazone (N=67) | Matching Placebo (N=71)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
Blood creatine phosphokinase increased (Investigations) | 12 | 9 | 11
Blood creatinine increased (Investigations) | 4 | 4 | 1
Blood urea increased (Investigations) | 5 | 1 | 0
Cataract (Eye disorders) | 4 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 3 | 3
Dizziness (Nervous system disorders) | 5 | 5 | 6
Fatigue (General disorders) | 8 | 2 | 3
Nausea (Gastrointestinal disorders) | 6 | 7 | 3
Oedema (General disorders) | 3 | 9 | 6
Protein urine present (Investigations) | 2 | 2 | 4
Proteinuria (Renal and urinary disorders) | 4 | 3 | 2
Tremor (Nervous system disorders) | 4 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 4
Urinary tract infection (Infections and infestations) | 2 | 3 | 4
Weight increased (Investigations) | 1 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No